CLINICAL TRIAL: NCT00937131
Title: A Study to Assess the Safety, Efficacy and Tolerability of Rituximab (Mabthera) in Combination With Plasma Exchange (PEX) in Patients With Acute Thrombotic Thrombocytopenic Purpura (TTP)
Brief Title: The Use of Rituximab in Acute Thrombotic Thrombocytopenic Purpura (TTP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/05/011
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no comparator (No Intervention)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Concentrate for solution for infusion, Intravenous use, 375mg/m2, Maximum 8 weekly infusions
  Other Names: Rituximab (MabThera)

SUMMARY:
TTP is a rare and serious blood disorder, characterized by the formation of small clots (micro thrombi) within the circulation and can be fatal. The formation of blood clots occurs primarily in the smaller blood vessels, the arterioles and capillaries, associated with multisystem organ involvement, especially the brain and kidneys. TTP has an incidence of approximately 1-3 people/million of the population/year.

TTP is due to a decrease in an enzyme, ADAMTS 13 that is released by cells lining blood vessels (endothelial cells). ADAMTS 13 'cleaves' or breaks down very large von Willebrand Factor (vWF) strands. vWF is used in blood clotting. Deficiency or inhibition of the enzyme, results in release of the ultra large vWF into the circulation. Platelets bind to these ultra large vWF multimers, promoting blood clot formation and platelet consumption (thrombocytopenia). In more then 70% of TTP cases no precipitating cause can be found and the majority of these patients have antibodies against ADAMTS 13. Plasma Exchange (PEX) was introduced in the management of TTP in 1977 and the mortality of TTP patients has since decreased from approximately 90% to 15-20%. PEX is essential in TTP treatment as plasma contains the missing enzyme ADAMTS 13.

Rituximab (licensed and internationally used monoclonal antibody) selectively acts on white blood cells known as B-lymphocytes or B cells that produce the antibody to ADAMTS 13. By inhibiting ADAMTS 13 antibody production, ADAMTS 13 activity increases, resulting in remission. Rituximab has been used in our institutions in patients with acute TTP that are refractory to standard treatment - PEX. The resulting remission has been dramatic, with a non-toxic side effect profile and no patients to date has relapsed (longest follow-up 19 months) following Rituximab therapy. Therefore, we plan to use Rituximab with PEX in patients who present with acute TTP.

DETAILED DESCRIPTION:
This is multi-centre study within the South East England (SEE) Thrombotic Thrombocytopenic Purpura (TTP) study group, primarily involving tertiary centres with expertise in treating TTP, apheresis units and specialist medical professionals. Feedback and discussions with TTP patients during treatment and discussion with those attending out-patient clinics have been incorporated into the development of this study. We have reviewed treatment protocols for TTP patients published in peer reviewed journals and consulted SEE TTP study groups on the study design. Medical professionals with expertise in TTP treatment and management have also been consulted.

This is a non-randomised Phase ll feasibility study to assess (i) whether Rituximab with PEX decreases the time to remission of patients with acute TTP, (ii) the mortality of TTP patients (assessed at 3 months from presentation), (iii) the safety and toxicity of Rituximab in conjunction with standard therapy for acute TTP, (iv) the effect of Rituximab on B cell function, (v) the effect of Rituximab on ADAMTS 13 activity and antibody production and time to relapse. The study design and methodology has been devised to specifically address questions regarding the use of Rituximab with PEX to further improve the treatment of TTP patients with the least disruption and inconvenience to their standard and local treatment and care to decrease TTP patient mortality.

Adult patients (across up to 8 participating UK sites) presenting with acute TTP and who fall within the study protocol inclusion criteria, as determined by the Lead Consultant Haematologist per institution, will be offered entry into the study. We wish to recruit 40 patients to this study and although the incidence of TTP is low, it is generally considered to be under diagnosed and therefore, underestimated. Recruiting 40 patients is achievable considering the number of patients presenting with acute TTP within the SEE TTP study group over the past 18 months. Some TTP patients may be unconscious or may have a neurological dysfunction associated with acute TTP, such as personality or memory symptoms. In these cases, consent will be requested from the patient's legal representative in compliance with the International Conference on Harmonisation (ICH) guidance for Good Clinical Practice (GCP).

Given the significant benefit in terms of remission, the increased level of ADAMTS 13 level in patients with acute refractory TTP and documented benefit of patients with other antibody driven disorders with Rituximab therapy, Rituximab in conjunction with standard therapy - PEX, is to be investigated. This is to reduce mortality further that the 15-20%, reducing the number of PEXs and therefore decreasing the exposure to blood component products that may contain fatal proteins such as variant Creutzfeldt-Jakob Disease (vCJD). As between 30-60% relapse with a further episode of TTP, follow up to determine time to relapse will be observed and compared to historical controls. During this period, blood counts and ADAMTS 13 levels will be assessed. We have a specific assay to determine the benefit following treatments and historical data to compare previous patient admission that can be matched. Researcher bias will be reduced as the time taken for a specific platelet level count (150 x 10 to the power of 9/L) must be determined and recorded within the routine laboratory in each institution, the number of PEX will be recorded by the patient's nurse, continuing until the platelet count is maintained above 150 x 10 to the power of 9/L. In addition, there will be a clear audit trail, which will allow data and records to be cross checked.

The investigators know from the literature and data collected as part of the SEE TTP study group, the epidemiology of TTP and mortality rate. With the improvement in laboratory techniques, there is improved detection of antibodies against ADAMTS 13. As antibodies to ADAMTS 13 can be detected in up to 90% of cases, having excluded specific precipitating causes, monitoring of ADAMTS 13 levels and the ADAMTS 13 antibody can be made regularly in our research facility. As per the patient's local treatment protocol for TTP i.e. PEX and steroid treatment, all patients will have a daily PEX until their platelet level count is > 150 X 10 to the power of 9/L. Patients will receive pre-Rituximab medication (Hydrocortison, Piriton, and Paracetamol, as per local protocol), 30 minutes prior to Rituximab infusion to reduce any potential side effects. Rituximab will be administered intravenously, immediately following PEX. PEX should be withheld for 24 hours following Rituximab therapy, if appropriate to the patient's clinical condition. Rituximab will be given once a week for 4 weeks in the first instance. The first treatment will be given within the first 3 days of admission, as there is a need to administer Rituximab in working office hours and allows participating sites to obtain the test results to ascertain whether the patient meets the study's inclusion criteria. If patients are well enough to be discharged before their 4th treatment, treatment will be continued in their local haematology day unit. If there is still evidence of antibodies to ADAMTS 13 and the ADAMTS 13 level has not been corrected/normalised, up to a maximum 4 additional Rituximab infusion will be given weekly. Nurses will monitor the patient's blood pressure, pulse, breathing rate, temperature and oxygen saturation level every 15 min for the first hour of Rituximab infusion and then hourly until infusion is complete. The patient will continue to be monitored as per the local protocol.

The side effects of Rituximab are generally mild such as flu-like symptoms, low blood pressure, nausea, flushing and rigor, and if experienced, usually occur during the first infusion. Pre-medication as noted above will be given prior to Rituximab infusion. If any side effects are experienced the rate of the infusion will be reviewed, slowed or suspended if necessary and intervention appropriate to the side effect will be given. Anaphylaxis is a potential risk with the first dose, but all patients will receive appropriate pre-medication. Very rare side effects are more likely to be associated with people who have extensive lymphoma disease and/or as a result of several years use of Rituximab in clinical trials, primarily for malignant disease, often with other chemotherapeutic agents as well as post marketing surveillance.

All patients will have standard haematological and biochemical blood tests as well having their ADAMTS 13 levels assessed. Regular blood tests will be arranged for patients discharged from hospital, to check their full blood count, electrolytes and liver function results and ADAMDTS 13 level. TTP patients will be reviewed initially weekly at their local out-patients clinic following discharge and as time passes and if their results are stable the period between appointments will be lengthened.

The study has been designed to cause the least disruption and inconvenience to patients and their standard and treatment/care. It is imperative that patients are continuously assessed and monitored during and post study treatment. Any potential risk is offset by (i) improving time to remission, associated with a decreased time of active TTP and organ damage, (ii) reduced exposure to plasma products and thus the risk of vCJD and (iii) improved management of acute TTP and mortality of these patients.

All patients will be reviewed in local haematology clinics or the TTP clinic at UCLH. Patients or their legal representatives will be informed or any update of TTP information in general or if new information becomes available about the treatment/drug during the study or during regular outpatient consultations. Review of ongoing data will be presented at the SEE TTP study group as well as national and international meetings. The final report will be presented in peer reviewed journals. Patient will also be kept informed of any publications arising from the study and hardcopies will be made available to all patients or their next of kin/legal representative.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years and < 65 years who present with an acute episode of TTP
* Evidence of microangiopathic haemolytic anaemia
* Thrombocytopenia with a normal clotting screen
* Raised Lactate Dehydrogenase (one and a half time above upper normal)
* Patients without neurological dysfunction able to give informed consent
* Patients of reproductive age (must avoid pregnancy for 12 months and/or normalised B cell function after receiving Rituximab. Oestrogen containing oral contraceptive pills and the morning after pills should be avoided in female TTP patients)
* Patients with an acute deterioration in neurological function which may include encephalopathy, such as altered personality, problems with short term memory and coma can be included when consent has been given by next of kin or from the appropriate legal representative.

Exclusion Criteria:

* All female subjects who are knowingly pregnant or breast feeding or do not use an adequate form of contraception (the effect on the foetus and newborn have not yet been fully established so Rituximab should be avoided in these groups. Male patients receiving Rituximab should ensure adequate contraception for 12 months following treatment).
* Patients who are HIV positive (which does not appear to be antibody mediated, would be unlikely to benefit from Rituximab)
* Patients with childhood TTP
* Patients who have Haemolytic Uraemic Syndrome (HUS) (which is not associated with reduced ADAMTS 13 levels)
* Patients who are post bone marrow transplant - either autologous or allogeneic
* Patients wiht a medical or long term psychiatric condition which, in the opinion of the investigator, contraindicates the patients' participation into the trial
* Previous or concurrent malignancies at other sites, with exception of appropriately treated localized epithelial or cervical cancer. Patients with a history of cured tumours may be entered (> 5 years).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate whether Rituximab and PEX decreases the time to remission of TTP patients. | One year

SECONDARY OUTCOMES:
Improved mortality ot TTP patients | 3 months
Safety and toxicity of Rituximab in conjunction with standard therapy for acute TTP | 3 months
Effect of Rituximab on B lymphocyte function | One year
Effect of Rituximab on ADAMTS 13 activity and antibody production and time to relapse | One year

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Scully, MBBS, BSc, MRCPath, Principal Investigator — University College London, University College London Hosptials NHS Trust
Locations (3):
- United Kingdom (3):
  - St Bartholomew's Hospital, London
  - St Thomas Hosptial, London
  - University College London Hospitals, London

REFERENCES:
- [Derived] Scully M, McDonald V, Cavenagh J, Hunt BJ, Longair I, Cohen H, Machin SJ. A phase 2 study of the safety and efficacy of rituximab with plasma exchange in acute acquired thrombotic thrombocytopenic purpura. Blood. 2011 Aug 18;118(7):1746-53. doi: 10.1182/blood-2011-03-341131. Epub 2011 Jun 2. PMID 21636861